CLINICAL TRIAL: NCT04410146
Title: The SQUID Trial for the Embolization of the Middle Meningeal Artery for Treatment of Chronic Subdural Hematoma (STEM)
Acronym: STEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balt USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIP-201912-SQUID
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Subdural Hematoma, Chronic
Keywords: Meningeal Arteries; Intracranial Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Hematoma, Subdural, Intracranial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Cognitive improvement, as measured by blinded assessment, utilizing the comprehensive neurocognitive battery.
  Imaging assessment by blinded core laboratory
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- SQUID (Experimental): Embolization of the Middle Meningeal Artery (MMA)
  Interventions: Device: SQUID Embolization; Device: SQUID Embolization and Surgical Evacuation
- No Embolization (Active Comparator): Standard Management
  Interventions: Procedure: Surgical Evacuation; Other: Other: Medical Management

INTERVENTIONS:
Device: SQUID Embolization — Embolization of the Middle Meningeal Artery using the SQUID non-adhesive liquid embolic agent
  Arms: SQUID
Device: SQUID Embolization and Surgical Evacuation — Embolization of the Middle Meningeal Artery using the SQUID non-adhesive liquid embolic agent and the surgical evacuation of the sub-dural hematoma
  Arms: SQUID
Procedure: Surgical Evacuation — Surgical evacuation of the sub-dural hematoma
  Arms: No Embolization
Other: Other: Medical Management — Standard
  Arms: No Embolization

SUMMARY:
STEM Study is a pivotal, international, multi-center, prospective, randomized (1:1) controlled trial designed to provide an assessment of the safety and effectiveness of Middle Meningeal Artery (MMA) embolization with SQUID for the management of Chronic Subdural Hematoma (cSDH)

DETAILED DESCRIPTION:
The study objective is to provide an assessment of the safety and effectiveness of Middle Meningeal Artery (MMA) embolization with SQUID for the management of Chronic Subdural Hematoma (cSDH).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Subject whose age is ≥ 30 at the time of consent
2. Pre-morbid mRS 0-1 within the previous 12 months
3. cSDH measures ≥ 10 mm in greatest thickness
4. cSDH exerts mass effect upon the subjacent brain, as indicated by local cortical flattening or midline shift
5. Imaging characteristics indicative of chronicity (≥ 50% of the volume of the collection should be isodense or hypodense to normal cortical gray matter on Computed Tomography (CT))
6. Subject presents with one or more of the following neurological symptoms: headache; cognitive decline; speech difficulty or aphasia; gait impairment or imbalance; focal neurological deficit (weakness, paresthesia or sensory deficit involving of one or more extremities or facial droop); and/or seizure
7. Subject, or his/her legally authorized representative, understands the nature of the procedure, consents to participation in the study and provides a signed Informed Consent Form
8. Female Subjects of child-bearing potential must be able to provide a current negative urine pregnancy test and agree to an appropriate method of contraception throughout the trial
9. Subject is able and willing to return to the investigational site for all follow-up visits (e.g., 30-day, 90-day, 180-day and 1-year), as required per protocol

Exclusion Criteria:

1. Subject with prior ipsilateral craniotomy or burr hole evacuation of cSDH
2. Subject with prior Embolization of either MMA
3. Subject requires (in the opinion of the treating surgeon) a full or mini craniotomy
4. Subject with urgent or emergent (within 1 hour of assessment) subdural hematoma evacuation needed
5. Subject with a cSDH with a focal location (confined to the frontal or temporal base or the inter-hemispheric space without cerebral convexity involvement)
6. cSDH developed due to underlying condition such as a vascular lesion, brain tumor, arachnoid cyst, spontaneous intracranial hypotension or secondary to a previous craniotomy
7. Life expectancy of <1 year
8. Subject who presents with an intracranial mass other than subdural hematoma
9. Subject who presents with a meningioma with mass effect and/or ≥1 cm or currently undergoing radiation therapy for carcinoma or sarcoma of the head or neck region
10. Subject with serum creatinine level > 3.0 mg/dL at time of enrollment (this will restrict the use of contrast) and not on dialysis
11. Subject with significant liver function impairment at the time of enrollment
12. Subject with a life-threatening allergy to radiographic contrast (unless treatment for allergy is tolerated or can be managed medically)
13. Subject who is currently enrolled in another investigational study protocol that could potentially confound the current study endpoints

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | On 180-day from intervention
  Treatment failure is defined by the occurrence of residual or re-accumulation of the SDH (≥10 mm) on 180-day scan from intervention.
Primary Effectiveness Endpoint | Within 180-days of intervention
  Treatment failure is defined by the occurrence of any of the following events:
  * Re-operation (after index procedure) or surgical rescue
  * Any new, major disabling stroke, myocardial infarction (MI) or death from any (neurological) cause
Primary Safety Endpoint | Within 30-days from intervention
  Major disabling stroke or any death

SECONDARY OUTCOMES:
mRS (analyzed as shift) | 180-day from intervention
Any investigational device/procedure-related AE/SAE | Through 1-year visit

OTHER OUTCOMES:
mRS (analyzed as shift) | 30-day and 1-year from intervention
mRS ≤ 2 (binary) | 30-day, 180-days, and 1-year from intervention
Cognitive improvement, as measured by blinded assessment, utilizing the comprehensive neuro-cognitive battery HVLT-R, COWAT, Animal Naming, Trail making tests | Baseline, 30-day, 180-day, and 1-year from intervention
EQ-5D-5L (including EQ-VAS) | Baseline vs. 30-day, 180-day, and 1-year from intervention
Hospital Days | Through 1-year visit
Intensive Care Unit (ICU) Days | Through 1-year visit
NIHSS | Baseline vs Discharge and 90-day
CT/MRI | Baseline vs. 180 days

CONTACTS AND LOCATIONS:
Overall Officials: David Fiorella, MD, PhD, Principal Investigator — Stony Brook University Medical Center; Adam Arthur, MD, MPH, Principal Investigator — Semmes-Murphy Neurologic and Spine Institute
Locations (32):
- United States (25):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Carondolet St. Joseph's, Tucson, Arizona
  - Riverside Community Hospital, Riverside, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - Swedish Medical Center, Englewood, Colorado
  - Baptist Health, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - University of Kansas, Kansas City, Kansas
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Nebraska Health, Omaha, Nebraska
  - Overlook Medical Center, Summit, New Jersey
  - NYU Langone Health, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Health Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Methodist University Hospital, Memphis, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Swedish Cherry Hill, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- France (4):
  - Chu Cote de Nacre, Caen
  - CHU Hopital Bicetre, Le Kremlin-Bicêtre
  - Hopital Pitie Salpetriere, Paris
  - CHU Hopital Maison Blanche, Reims
- Germany (2):
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum Nurnberg Sud, Nuremberg
- Gregorio Maranon Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fiorella D, Monteith SJ, Hanel R, Atchie B, Boo S, McTaggart RA, Zauner A, Tjoumakaris S, Barbier C, Benitez R, Spelle L, Pierot L, Hirsch JA, Froehler M, Arthur AS; STEM Investigators. Embolization of the Middle Meningeal Artery for Chronic Subdural Hematoma. N Engl J Med. 2025 Feb 27;392(9):855-864. doi: 10.1056/NEJMoa2409845. Epub 2024 Nov 20. PMID 39565980